CLINICAL TRIAL: NCT04376463
Title: Effects of a Multicomponent Exercise and Supplementation of Branched Chain Aminoacids Health Parameters in the Dwelling Elderly
Brief Title: Effects of a Multicomponent Exercise and Supplementation of BCAA´s in Immunity System Dwelling Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Adriana Caldo, Researcher, principal investigator, University of Coimbra
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UC
Record Dates: First submitted 2020-04-13; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Frail Elderly Syndrome; Physical Exercise
Keywords: Branched Chain Aminoacids Supplementation; Frail Elderly; Dwelling Elderly; Multicomponent Exercise; Immunology
MeSH Terms: conditions — Motor Activity | interventions — Amino Acids; Exercise

STUDY DESIGN:
Intervention Model Description: It was an experimental design, controlled, non-randomized, with a convenience sample of 16-week supplementation combined or not with exercise. All participants in the groups ME+BCAA and BCAA received at the beginning of the protocol a bottle with assigned codes with flavourless powder (BCAA), and a dosage of 0.21g/kg/session. They took the supplement with 200 ml of water immediate after exercise, in the ME+BCAA group, and at the same time in the BCAA group (Ispoglou et al., 2016). Throughout the intervention period, all tests and intervention were done after breakfast and before lunch (supplementation, physical exercise, data collection, questionnaires, physical tests), and 30-60 minutes before lunch. The ME group just folowed the exercice protocol, and CGne group did not alter their usual routine.
Who Masked: Investigator
Masking Description: It is an experimental design, controlled with 8 months of supplementation combined with exercise and washout 2 months, totalling 10 month intevention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mood state and aminoacids supplementation (Experimental): The aim of this study was to analyse the isolated and combined effects of BCAA supplementation and exercise on physical frailty status and mood states in pre-frail institutionalized older women.
  Interventions: Dietary Supplement: Branched Chain Aminoacid
- Physical Tests (Experimental): Through the combination of bcaa supplementation and physical exercise is able to improve the functional capacity of the elderly, through the SPPB test battery, short performance physical battery.
  Interventions: Dietary Supplement: Branched Chain Aminoacid
- Psychometrics evaluated (Experimental): Through the combination of bcaa supplementation and physical exercise, it is able to improve moods and cognition of the elderly.
  Interventions: Dietary Supplement: Branched Chain Aminoacid
- Fried Scale Phenotype (Experimental): Primary outcomes include Physical Frailty evaluated according to Fried's Frailty Phenotype2): Shrinking assessed by self-report of unintentional weight loss of four kilograms or more in the last six months; Self-reported exhaustion evaluated by concordance of two questions (7 and 20) of the Center for Epidemiology-Depression (CES-D) scale; Weakness analyzed using the handgrip strength test; Slowness measured by the 4.6 meters walking test; levels of Physical Activity assessed by the (IPAQ).
  Interventions: Dietary Supplement: Branched Chain Aminoacid

INTERVENTIONS:
Dietary Supplement: Branched Chain Aminoacid — It is an experimental design, controlled with 8 months of supplementation combined with exercise and washout 2 months, totalling 10 month intervention.
  Other Names: Physical Exercise

SUMMARY:
The frailty syndrome (FS) is characterized by a multifactorial clinical syndrome, which includes 5 items, 1 - Change in body composition, 2 - Holding force, 3 - Fatigue reported, 4 - Reduction of walking speed, 5 - Low physical activity. The cumulative effect of deficits on the physiological functions caused by the syndrome results in early physical and cognitive loss. It is known that physical exercise, associated with protein supplementation are examples of non-pharmacological treatments that can promote functional and structural adaptive responses of the skeletal muscle system. One of the factors related to frailty is the reduction of body and muscle mass. Branched-chain amino acids, especially leucine, are nutrients that influence the adaptative response of muscle. It is intended through a physical exercise program (multicomponent = exercise of strength + aerobic exercise), to attenuate the effects of ageing and mainly of physical and cognitive frailty, evaluating the health parameters of frail elderly, alone or together with supplementation (BCAA), branched-chain amino acids, modulation of immune markers, markers of malnutrition and the skeletal muscle system in frail and pre-frail dwelling elderly people living in the city of Coimbra. To achieve that, the following parameters will be evaluated: biosocial indicators, anthropometric evaluation and body composition, indicators of global health and functional physical fitness, inflammatory biomarkers, neuroendocrine, signs of skeletal muscle function, evaluation of quality of life related to emotional state, cognitive profile and frailty-trait evaluation. The results obtained from the indicators, markers and questionnaires used are expected to contribute to the attenuation of frailty, improving the health and quality of life of the elderly.

Keywords: frail elderly, multicomponent exercise, branched chain amino acid, healthy life

DETAILED DESCRIPTION:
This investigation was conducted in accordance with the guidelines laid down in the Declaration of Helsinki. All procedures were approved by the University Faculty Research Ethics Committee and written informed consent was obtained from all participants. This PhD project is inserted in the thematic line of the (CIDAF) Research Centre in Physical Activity and Ageing; Ageing: Is It Ever Too Late to be Active and Healthy / Fit? This project will also be sent to the homes of all the participants in the study to sign a term so that they can sign a consent for the implementation of the study at their premises.

During the period of the intervention of the exercise and after the experimental period, an interview will be done through questionnaires, biosocial and overall health status. The main results will be the cognitive, biosocial and overall health status. There will be a session to administer a test battery on the overall health status, cognitive status (screening of cognition), and screening for mobility. Secondary measures include psychological well-being, cognition, anthropometric, immunological, and neurological parameters.

Experimental design (supplementation time)

It is an experimental design, controlled with 6 months of supplementation combined with exercise. Participants will receive a code number according to the order of recruitment. The participants sample was non-randomization, sample was convenience, will be performed using the assignment list and code number after recruitment for the study. Initially the elderly will be divided into 4 groups: Multicomponent Exercise + BCAA (ME+BCAA) group 1, Multicomponent Exercise (ME) group 2, BCAA group 3, Control non-exercise (CONTROL) group 4. Data collection was performed at 4 moments,1-Initial time (baseline), 2-After 16 weeks training period, 3-After 8 weeks detraining period and 4-After 16 weeks period, totaling 4 collections throughout the project and 40 weeks.

The supplement was supplied through the company and has about 95% purity and trade certification in the EU. The subjects ingested 1 sachet (0,21g/kg/session) prepared after to finish exercise by mixing the contents of each sachet with 200mL water and consuming as follows: first beverage during the morning after breakfast and before lunch.

ELIGIBILITY:
Inclusion Criteria:

* Fried criteria

Exclusion Criteria:

* Dementia
* Morbid obesity, and the use of medications that may cause great attention impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-13 (Actual); Primary Completion 2019-09-14 (Actual); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
THE INDEPENDENT AND COMBINED EFFECTS OF A 16-WEEK EXERCISE AND BCAA SUPPLEMENTATION ON FRAILTY MARKERS AND MOOD STATES OF OLDER WOMEN | up to 24 weeks
  Physical function and muscle strength Short physical performance battery (SPPB) was used to assess gait speed, chair stand, and balance tests. This SPPB test is composed of 3 subdimensions: i) static balance (composed of 3 tests), ii) muscular strength of the lower limb, which consist of get up and seat in a chair, 5 times, with arms crossed at the chest, and iii) 3-meter test, that marks the time to travels the 3-meter course, in the usual speed (Guralnik et al., 1994).
Geriatric Depression Scale | up to 24 weeks
  The GDS-15, (Yesavage, 1982) consisting of 15 direct questions with yes or no answers, which evaluate e classify the psychological condition related to depression and its symptoms. The score result has 3 response modes 0 to 5 points indicates normal psychological condition, (no symptoms of depression), 6 to 10 points indicates (mild depressive symptoms), 11 to 15 indicates (symptoms of serious depression). The scale GDS was translate in Portuguese by (Apóstolo, 2014).

SECONDARY OUTCOMES:
Profile of Mood State short version (POMS-sv) | through study completion, an average of 1 year
  Profile of Mood State (McNair, 1971) is a test to evaluated individual's mood state. This tool, self-related and easy to use, is able to verify a transient profile. A short version (Raglin & Morgan, 1989) was applied to facilitate use. POMS consist of 22 Likert-type question, divided in six dimensions with scales from 0 to 4. The final score consists of a sum of all negative dimensions subtracting the positive dimension of Vigour. Total Mood Disturbance (TMD) scores of Profile of Mood States (T+D+H+F+C)-V), (Tension-anxiety, depression-melancholia, Hostility-anger, Fatigue-inertia, Confusion, and Vigour), (Viana, Almeida, & Santos, 2001).
Mini Nutritional Assessment | through study completion, an average of 1 year questionnaire of nutrition
  Mini Nutritional Assessment The Mini Nutritional Assessment is calculated with a maximum total score of 30 points, in which the result of 17 points and below is characterized as malnourished, between 17 to 23.5 points, indicates a risk of malnutrition, and a score above 23.5 is normal nutritional status. A normal nutritional status was used to evaluate the nutritional status and the participants were classified as: Total points in the MNA® evaluation section (maximum 16 points). The results found will be sent to a nutritionist, (Loureiro, 2008). All participants were provided with similar diets, in terms of caloric intake and nutrients, controlled by a local nutritionist during the intervention period.
The Charlson Comorbidity Index | through study completion, an average of 1 year (questionnaire) physiological parameter
  The Charlson comorbidity index was used to classify comorbid conditions based on the registry of each individual comorbidity and was combined with age and gender to form a single index (Charlson et al., 1987).

CONTACTS AND LOCATIONS:
Locations (1):
- Adriana Caldo, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No
This is a controlled longitudinal study experimental design, with 8 months of supplementation combined with exercise and washout 2 months, totalling 10 months intervention. Participants will receive a code number according to the order of recruitment. Initially the elderly will be divided into 4 groups: Multicomponent Exercise + BCAA (ME+BCAA) group 1, Multicomponent Exercise (ME) group 2, (BCAA) group 3, Control non-exercise (CONTROL) group 4. The collection of data for the different variables will be 1-baseline, 2-post intervention (after 4 months of intervention), 3-washout period (after 2 months "detraining"), 4-final period (after 4 months intervention).